CLINICAL TRIAL: NCT02599532
Title: Pharmacokinetics of Apixaban in Nephrotic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-1455; 550KR161709 (Other Grant/Funding Number: NCTraCS)
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Nephrotic Syndrome; Proteinuria
Keywords: Apixaban; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nephrotic syndrome (Other): Subjects with nephrotic syndrome will receive a single dose of apixaban 10 mg and will subsequently have blood drawn at 0, 0.5, 1, 3, 4, 6, 8, 24 hours after drug administration.
  Interventions: Drug: apixaban
- Non-nephrotic syndrome (Other): Subjects without nephrotic syndrome will receive a single dose of apixaban 10 mg and will subsequently have blood drawn at 0, 0.5, 1, 3, 4, 6, 8, 24 hours after drug administration.
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: apixaban — Study subjects will be given a single-dose of apixaban 10 mg.
  Other Names: Eliquis

SUMMARY:
This study is to investigate the pharmacokinetics and pharmacodynamics of apixaban in nephrotic syndrome.

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is characterized by proteinuria and hypoalbuminemia, and patients with nephrotic syndrome are known to be hypercoaguable with increased incidence of venous thromboembolism necessitating anticoagulation. While classically warfarin has been used as an anticoagulant in NS, newer oral anticoagulants, such as apixaban, are increasingly used to treat venous thromboembolism (VTE) in the general population. It is unknown how hypoalbuminemia and proteinuria affect the pharmacokinetics and pharmacodynamics of apixaban.

This will be a parallel arm, single-dose pilot study of the pharmacokinetics of apixaban in adults with nephrotic syndrome. Goal enrollment of twenty subjects with non-diabetic nephropathy who have nephrotic-range proteinuria, defined as >3.5g/24 hours or UPC >3.5 and ten healthy control subjects without nephrotic syndrome. Each subject will be administered a single dose of apixaban 10 mg. Plasma drug concentration level and plasma anti-Xa activity levels will be measured at 0, 0.5, 1, 3, 4, 6, 8, 24 hours after drug administration in order to determine the maximum plasma concentration of apixaban, area under the curve, and half-life of apixaban in the setting of hypoalbuminemia and proteinuria due to nephrotic syndrome. Apixaban levels will be measured via liquid-chromatography spectrometry mass. Additionally, thrombin generation will be measured at 0, 3, 6, and 24 hours.

ELIGIBILITY:
* Inclusion Criteria:

  * Study subjects:

    * Between 18 and 79 years old
    * Confirmed diagnosis of Nephrotic Syndrome, with at least one of the following:

      * 1. Nephrotic-range proteinuria, defined as >3.5 g/24 hours or UPC >3.5 (confirmed within 1 month prior to scheduled study visit)
      * 2. Hypoalbuminemia, defined as <3 g/dL (confirmed within 1 month prior to scheduled study visit)
  * Control subjects:

    * Between 18 and 79 years old
    * Normal albumin levels (≥3.5 mg/dL)
    * No proteinuria (UPC <0.15)
* Exclusion criteria:

  * Age <18 or ≥ 80 years old
  * SCr ≥ 1.5 AND weight ≤ 60kg (these subjects would receive a reduce dose of apixaban, per drug labeling)
  * On dialysis
  * Baseline prolonged PT/INR, PTT (as defined by greater than the upper limit of normal)

    * INR will be used as the primary lab value to evaluate bleeding risk (e.g. a patient presenting with an INR within normal limits, but prolonged PT or PTT, will not meet this exclusion criterion and will still be eligible for the study)
    * Reference Ranges

      * INR: >1.4
      * PT: >13.3 sec
      * aPTT: >37.7 sec
  * Platelets <100
  * History of GI bleed
  * History of intracranial bleed
  * History of stroke
  * Use of (but not limited to) the following medications within the past 14 days:

    * Inducers of CYP3A4 (e.g. rifampin, carbamazepine, phenytoin, St. John's wort, etc.)
    * Strong inhibitors of CYP3A4 (e.g. ketoconazole, ritonavir, clarithromycin, etc.)
    * Antiplatelet and/ or anticoagulant agents: heparin, aspirin* (see below), clopidogrel, prasugrel, NSAIDs, warfarin, rivaroxaban, dabigatran, edoxaban
    * Selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitors (SNRI)
  * Pregnancy/breastfeeding
  * Liver disease with impaired synthetic function (INR >1.4, total bilirubin >1.2)
  * Congestive heart failure

Special consideration for patients on aspirin: for patients on chronic low-dose aspirin therapy, we will allow a 7 day wash out period. This will only be allowed for patients who are taking aspirin as primary prophylaxis or for unclear indications. Patients who are on aspirin therapy for following indications will be excluded: primary prophylaxis of stroke due to atrial fibrillation, secondary prevention of stroke or myocardial infarction, history of coronary artery disease or peripheral vascular disease. For patients who meet the potential criteria for the 7-day wash out, their medical history will be reviewed by one of the clinician investigators to ensure that it is safe and appropriate to hold the agent.

Those subjects taking aspirin for the following reasons will be excluded:

* Primary stroke prevention from atrial fibrillation
* Secondary prevention due to prior stroke, heart attack or cardiac stent
* Existing heart disease or peripheral vascular disease.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve after single dose (AUC) of apixaban | Predose; 0.5, 1, 3, 4, 6, and 8 hours (hr) postdose on Day 1; 24 hours postdose on Day 2

SECONDARY OUTCOMES:
Mean terminal phase plasma half-life (t½) | Predose; 0.5, 1, 3, 4, 6, and 8 hours postdose on Day 1; 24 hours postdose on Day 2
Apparent oral clearance (CL/F) | Predose; 0.5, 1, 3, 4, 6, and 8 hours postdose on Day 1; 24 hours postdose on Day 2
Maximum observed drug concentration in plasma after single dose administration (Cmax) | Predose; 0.5, 1, 3, 4, 6, and 8 hours postdose on Day 1; 24 hours postdose on Day 2
Thrombin Generation Assay | Predose; 3 and 6 hours postdose on Day 1; 24 hours postdose on Day 2
Anti-Xa activity | Predose; 0.5, 1, 3, 4, 6, and 8 hours postdose on Day 1; 24 hours postdose on Day 2

OTHER OUTCOMES:
Proportion of germline variants in genes involved in apixaban metabolism and clearance | DNA extracted from whole blood specimens will be genotyped at the conclusion of enrollment, approximately 12 months.
  Explore the relationship between variant genes responsible for apixaban metabolism and clearance (CYP3A4/5, CYP1A2, CYP2J2, ABCB1, and ABCG2) and drug exposure as measured by AUC. Genotyping analyses will be performed at conclusion of study and appropriate conventional statistical analyses will be employed to assess all genotype-phenotype associations.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Crona, PharmD, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Vimal Derebail, MD, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States